CLINICAL TRIAL: NCT05886673
Title: Development of a Protective Cream Against Radiodermatitis Caused by Radiotherapy.
Acronym: RADIOCREMVAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Antonio J. Conde Moreno (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Sponsor-Investigator, Antonio J. Conde Moreno, Investigator, Instituto de Investigacion Sanitaria La Fe
Organization: Instituto de Investigacion Sanitaria La Fe (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-963-1
Record Dates: First submitted 2023-05-11; First posted 2023-06-02 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Radiodermatitis
Keywords: radiodermatitis; oncology; radiotherapeutic oncology
MeSH Terms: conditions — Radiodermatitis; Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study treatment (Experimental): The experimental cream formulation has the same components as the control plus 2% pterostilbene, 1% silibinin and 2% nicotinamide riboside.
  Interventions: Other: experimental cream
- Control treatment (Other): The control cream formulation is designed to help maintaining skin hydration and texture. It contains common ingredients largely used in cosmetics: stearic acid, cetyl alcohol, liquid vaselin, isopropyl myristate, triethanolamine, methyl paraben, propyl paraben, propylene glycol, ethoxydiglycol, and water.
  Interventions: Other: standard of care

INTERVENTIONS:
Other: experimental cream — experimental cream
  Arms: Study treatment
Other: standard of care — standard of care
  Arms: Control treatment

SUMMARY:
The study cream is to be evaluated in a multicenter, randomized, controlled clinical study carried out in 2 hospitals, in the Radiation Oncology service of Valencia to evaluate its radioprotective and radiomitigation effect in the prophylactic treatment of acute radiodermatitis caused by radiation.

A total of 82 patients with squamous cell carcinoma of the head and neck (SCCHN) were are going to be randomized in a study. Patients receive the study topical cream or "standard" skin care from Hospitals where the study is carried out. All patients will be treated with a combination of fractionated radiotherapy and platinum-based chemotherapy OR cetuximab for curative purposes.

The main objective of the study cream is to obtain a reduction in the number of patients who experience acute radiation dermatitis grade 3 or 4 (NCI CTCAE version 4.03) to grade 2, the last day of treatment. As a secondary objective, to obtain a reduction in the number of patients experiencing grade 3 or 4 to grade 0 acute radiation dermatitis, within a month of finish treatment. All patients will be evaluated periodically. The skin is photographed irradiated and all changes of radiation dermatitis are classified. The valuation of the radiodermatitis will be carried out objectively using a thermograph. In addition, the patients who complete questionnaires about their quality of life (QLQ-C30). These Questionnaires are answered in weeks 1, 2, 3 and 4 of treatment, as well as at the end of the radiation therapy or chemotherapy.

For the primary endpoint of radiodermatitis with CTCAE ≥ grade 2, assessments are made according to the protocol (PP), in addition to the primary intention-to-treat (ITT) approach. In this PP analysis, the patients are excluded according to protocol definition or meeting decisions preanalysis, respectively. The study is designed as a randomized trial with a 1:1 allocation to the two groups.

The secondary objective is to study a reduction in the percentage of patients experiencing radiation dermatitis with a maximum CTCAE grade 3 or 4 during the period of treatment and in the follow-up period of one month, thanks to the application of the cream of study.

DETAILED DESCRIPTION:
The study will be a randomized, controlled, parallel, prospective, double-blind, two-armed clinical study with a cosmeceutical product.

The creams (experimental cream (CE) and standard of care (SC)) will be randomly distributed among the patients, so that 50% receive CE and the other 50% SC. Each tube will have a number whose content does not neither the evaluators and the patients will know.

In a period between January 2023 and June 2023, the radiation oncology services of Hospitals La Fe and Clinic de Valencia conducted a study on 82 patients with SCCHN. what will they be undergoing external beam radiotherapy with or without concomitant chemotherapy.

Radiotherapy treatment uses techniques of modulated intensity of the radiation beam (IMRT or VMAT) image-guided (IGRT) that offer very high precision in the daily administration of treatment, improving the tolerance of healthy tissues and the quality life of patients.

Patients will be divided into two groups:

Group A (intervention, CE): this group will receive the topical application of the study cream.

Group B (control, SC): standard care will be applied to this group.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed localized (nonmetastatic) SCCHN.
* 18 years or older, with ECOG (Eastern Cooperative Oncology Group) Performance Status of performance from 0 to 2, a life expectancy of 6 months or more, and with signed informed consent.
* Intact skin at the start of radiotherapy.

Exclusion Criteria:

* Distant metastases, prior radiation therapy for SCCHN.
* Ongoing participation in any other study or clinical trial.
* Pregnant or lactating.
* Hypersensitivity to any of the components of the study cream.
* Prior or concurrent cancer within 5 years of study start and any other social or medical condition that may affect participation in or evaluation of the study will be excluded.
* History of collagen disease, such as systemic lupus erythematosus and/or scleroderma.
* Present dermatological conditions, such as psoriasis, bullous pemphigus or epidermolysis bullosa or bullosa.
* Inflammatory changes in the skin of the area to be irradiated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Reduction the occurrence of grade 2 radiodermatitis | Through study completion, an average of 4 months
  Reduction (in the progression to severe radiation dermatitis) of the number of patients experiencing acute radiation dermatitis from grade 3 or 4 to grade 2 on the last day of treatment.
Delay in the occurrence of grade 2 radiodermatitis compared to the placebo group. | Through study completion, an average of 4 months
  Delay in the occurrence of grade 2 radiodermatitis compared to the placebo group.

SECONDARY OUTCOMES:
Incidence of radiodermatitis | through study completion, an average of 4 months
  To compare the percentage of patients (incidence) with radiodermatitis, the degree of toxicity and the percentage of cases with radiodermatitis grade 2 or higher in patients undergoing the different treatments, in the total sample and stratified by number of radiotherapy sessions per month and at the end of treatment.
  To assess and compare the time to onset of each grade of skin reaction; to identify the frequency and location of specific features of radiodermatitis.
  To study the health-related quality of life perceived by patients at the beginning and at the end of radiotherapy. of radiotherapy. To evaluate and compare the local symptoms described by patients during radiotherapy treatment and treatment and assessed by PREMS-PROMS.
  To compare the temperature of the irradiated area using a thermograph during radiotherapy, in the 4 visits to be made by the patient. the 4 visits to be made by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio J Conde Moreno, Principal Investigator — Medical Research Institut La Fe
Locations (1):
- Medical Reserarch Institute La Fe, Valencia, Spain

DOCUMENTS (2):
  • Study Protocol (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT05886673/Prot_000.pdf
  • Informed Consent Form (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT05886673/ICF_001.pdf